CLINICAL TRIAL: NCT00646113
Title: An Open, Prospective, Single Arm, Multi-centre Study Evaluating OsseoSpeed™ Implant 3 mm Diameter Replacing a Central or Lateral Mandibular Incisor or Lateral Maxillary Incisor. A 5-year Follow-up Study.
Brief Title: Study Evaluating OsseoSpeed™ Narrow Implant in the Upper and Lower Anterior Jaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-NAR-0001
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OsseoSpeed™ TX 3.0S (Dental implant) (Experimental): OsseoSpeed™ TX 3.0S, Dental implants, 3.0 mm diameter, in lengths of 11, 13 and 15 mm
  Interventions: Device: OsseoSpeed™ TX 3.0S

INTERVENTIONS:
Device: OsseoSpeed™ TX 3.0S — OsseoSpeed™ TX 3.0 mm diameter

SUMMARY:
To evaluate 5-year survival, functionality and safety for OsseoSpeed™ 3.0 mm diameter implant when used for single tooth crown in positions 12, 22, 31, 32, 41 and 42. The primary hypothesis is that implant survival after 5 years is equal to what has been observed with comparable implants in current literature.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Aged 18-70 years at enrolment
* History of edentulism in the study area of at least two months
* Presence of natural tooth roots adjacent to the study implant position
* Deemed by the investigator to have a bone height and width suitable for 3.0 mm diameter study implant
* Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

* Unlikely to be able to comply with study procedures, as judged by the investigator
* Uncontrolled pathologic processes in the oral cavity
* Known or suspected current malignancy
* History of radiation therapy in the head and neck region
* History of chemotherapy within 5 years prior to surgery
* Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration, as deemed by the investigator
* Uncontrolled diabetes mellitus
* Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
* Smoking more than 10 cigarettes per day
* Present alcohol and/or drug abuse
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
* Previous enrolment in the present study
* Simultaneous participation in another clinical study, or participation in a clinical study during the last weeks prior to enrolment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo Moreno, Assoc. Prof., Principal Investigator — University of Granada: School of Dentistry
Locations (6):
- Tand-mund-kaebekirurgisk Klinik, Copenhagen, Denmark
- Bundeswehrkrankenhaus, Ulm, Germany
- Clinica Odontoiatrica, Milan, Italy
- Department Oral Surgery, University of Granada: School of Dentistry, Granada, Spain
- Käkkirurgiska kliniken, Odontologiska Institutionen, Jönköping, Sweden
- Bristol Dental Hospital and School, Bristol, United Kingdom

REFERENCES:
- [Result] Galindo-Moreno P, Nilsson P, King P, Becktor J, Speroni S, Schramm A, Maiorana C. Clinical and radiographic evaluation of early loaded narrow diameter implants - 1-year follow-up. Clin Oral Implants Res. 2012 May;23(5):609-16. doi: 10.1111/j.1600-0501.2011.02254.x. Epub 2011 Sep 28. PMID 22093047
- [Result] Maiorana C, King P, Quaas S, Sondell K, Worsaae N, Galindo-Moreno P. Clinical and radiographic evaluation of early loaded narrow-diameter implants: 3 years follow-up. Clin Oral Implants Res. 2015;26(1):77-82. doi: 10.1111/clr.12281. Epub 2013 Oct 30. PMID 25650268
- [Result] King P, Maiorana C, Luthardt RG, Sondell K, Oland J, Galindo-Moreno P, Nilsson P. Clinical and Radiographic Evaluation of a Small-Diameter Dental Implant Used for the Restoration of Patients with Permanent Tooth Agenesis (Hypodontia) in the Maxillary Lateral Incisor and Mandibular Incisor Regions: A 36-Month Follow-Up. Int J Prosthodont. 2016 Mar-Apr;29(2):147-53. doi: 10.11607/ijp.4444. PMID 26929953
- [Result] Galindo-Moreno P, Nilsson P, King P, Worsaae N, Schramm A, Padial-Molina M, Maiorana C. Clinical and radiographic evaluation of early loaded narrow-diameter implants: 5-year follow-up of a multicenter prospective clinical study. Clin Oral Implants Res. 2017 Dec;28(12):1584-1591. doi: 10.1111/clr.13029. Epub 2017 Jun 18. PMID 28626888

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- OsseoSpeed™ TX 3.0: OsseoSpeed™ TX 3.0 mm diameter implants (lengths 11 mm, 13 mm and 15 mm).
Period: Overall Study
Arm/Group | OsseoSpeed™ TX 3.0
Started (Completed surgery) | 69; 97 Implants (3 of the 72 enrolled participants were excluded before surgery.)
Completed | 61; 86 Implants
Not Completed | 8; 11 Implants
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Number of enrolled participants that completed surgery (Baseline)
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX 3.0S
Number analyzed (Participants) | 69
Number analyzed (Implants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 36
Region of Enrollment [Number; unit: participants]
  Sweden | 15
  Denmark | 14
  United Kingdom | 12
  Italy | 10
  Germany | 4
  Spain | 14

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: Overall implant survival rate evaluated clinically and radiographically
Time Frame: Evaluated at implant placement and at the 5 years follow-up after implant placement
Population: A total of 69 subjects were enrolled in the study and received a total of 97 implants.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Groups:
- OsseoSpeed™: OsseoSpeed™ TX 3.0 mm diameter
Arm/Group | OsseoSpeed™
Number analyzed (Participants) | 69
Number analyzed (Implants) | 97
Implants | 93

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | OsseoSpeed™ TX 3.0S
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 39/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed™ TX 3.0S (N=69)
Crown loss (Product Issues) | 10 (10) — 10 subjects experienced temporary crown loss. Resolved by having the crowns re-cemented.
Abutment fractures (Product Issues) | 7 (7) — 7 subjects experienced implant abutment fractures
Implant lost (Product Issues) | 4 (4) — 4 participants lost their implants. 3 due to insufficient osseointegration and 1 due to infection. All 4 implants were lost during the healing phase before loading of the implant.
Common cold (Infections and infestations) | 14 (30)
Headache (General disorders) | 4 (8) — Headache and/or Migraine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less